CLINICAL TRIAL: NCT01996943
Title: Investigating the Effects of Ethanol on Atrial Fibrillation Susceptibility and Pathogenesis
Brief Title: The HOLIDAY (HOw ALcohol InDuces Atrial TachYarrhythmias) Study
Acronym: HOLIDAY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 12-08579; 1R01AA022222-01 (NIH)
Record Dates: First submitted 2013-09-30; First posted 2013-11-27 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Atrial Fibrillation; Alcohol
Keywords: Atrial Fibrillation; Alcohol; Electrophysiologic properties of the atria; Randomized Clinical Study
MeSH Terms: conditions — Atrial Fibrillation | interventions — Ethanol; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): The placebo will be administered to participants after the baseline electrophysiologic measurements are recorded.
  Interventions: Drug: Placebo
- Ethanol (Active Comparator): Ethanol (alcohol) will be administered to participants after the baseline electrophysiologic measurements are recorded.
  Interventions: Drug: Ethanol

INTERVENTIONS:
Drug: Ethanol — 6% volume/volume ethanol in 0.45% saline solution.
  Other Names: Alcohol
  Arms: Ethanol
Drug: Placebo — The placebo with be 0.45% saline solution ("half normal saline").
  Other Names: Saline
  Arms: Placebo

SUMMARY:
Atrial fibrillation (AF) is the most common sustained arrhythmia in the United States and it has been associated with ethanol use. Understanding how ethanol affects the electrical properties of the heart and induces AF has important public health implications. The objective of this research is to investigate the mechanistic relationship between ethanol and atrial fibrillation in humans by performing a placebo controlled study looking at the electrical properties of the heart in patients receiving intravenous ethanol or placebo. The investigators hypothesize that ethanol increases the susceptibility of human myocardium to atrial fibrillation through electrophysiologic changes in the atrial myocardium in the acute setting.

DETAILED DESCRIPTION:
The purpose of this study is to look for changes in the electrical properties of heart that may be caused by ethanol (commonly referred to as alcohol) and specifically how ethanol may trigger episodes of the most common abnormal heart rhythm, atrial fibrillation (AF). This study will demonstrate the mechanism of ethanol induced atrial fibrillation and clarify the health effects of one of the worlds' most popular drugs (ethanol). With this understanding, physicians may be able to better identify those patients most at risk for ethanol induced AF and target public health campaigns towards this vulnerable population.

Patients in this study will undergo an electrophysiologic study both prior to and after receiving either an ethanol or placebo infusion. This electrophysiology study will measure AF inducibility (the primary outcome), left and right atrial conduction times, and the atrial effective refractory period in multiple locations (AERP). The changes in the conduction times and AERPs (before and after study drug infusion) will be recorded as secondary outcomes.

About 100 people will participate in this study. 50 people will be randomized to receive intravenous ethanol, and 50 people will be randomized to receive an intravenous placebo. The placebo will be in the form of 0.45% saline solution ("half normal saline") and the alcohol will be in the form of 6% volume/volume ethanol in 0.45% saline solution.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21-80 with paroxysmal atrial fibrillation (AF), supraventricular tachycardia, or undifferentiated palpitations who are to undergo either an elective ablation procedure (for AF, atrial flutter, atria tachycardia, atrial ventricular nodal reentrant tachycardia (AVNRT), or atrial ventricular reentrant tachycardia (AVRT)) or a diagnostic electrophysiology study in order to diagnose and treat their clinical arrhythmia at the University of California, San Francisco (UCSF) will be eligible for enrollment.

Exclusion criteria:

* Patients will be excluded if they are not in normal sinus rhythm (i.e. in AF, atrial tachycardia, atrial flutter, or incessant AVNRT/AVRT) at the time of onset of the procedure, any history of substance abuse or alcoholism as determined by history, AUDIT questionnaire, or chart review, left ventricular ejection fraction <50%, inability to give informed consent, liver dysfunction (elevated aspartate aminotransferase , alanine aminotransferase, total bilirubin, or alkaline phosphatase >2x normal), clinical evidence of liver disease (enlarged liver, caput medusa, spider angiomas, or other signs of liver disease on exam), or pregnancy.

Ages: 21 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2019-05 (Actual); Study Completion 2020-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory M Marcus, MD, MAS, Principal Investigator — University of California, San Francisco; Jonathan W Dukes, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Result] Marcus GM, Dukes JW, Vittinghoff E, Nah G, Badhwar N, Moss JD, Lee RJ, Lee BK, Tseng ZH, Walters TE, Vedantham V, Gladstone R, Fan S, Lee E, Fang C, Ogomori K, Hue T, Olgin JE, Scheinman MM, Hsia H, Ramchandani VA, Gerstenfeld EP. A Randomized, Double-Blind, Placebo-Controlled Trial of Intravenous Alcohol to Assess Changes in Atrial Electrophysiology. JACC Clin Electrophysiol. 2021 May;7(5):662-670. doi: 10.1016/j.jacep.2020.11.026. Epub 2021 Jan 27. PMID 33516710

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Ethanol
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ethanol | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 28 | 34 | 62
  >=65 years | 22 | 16 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.14 (13.08) | 58.78 (11.27) | 60.51 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 38 | 36 | 74
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 50 | 48 | 98
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 45 | 44 | 89
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Atrial Fibrillation Induction
Description: Induction of Atrial fibrillation will be attempted by pacing and isoproterenol infusion following study drug infusion. The ability to induce atrial fibrillation (yes or no) will be recorded as the primary outcome.
Time Frame: This will be measured after study drug (ethanol or placebo) infusion. The measurement will be performed within 1 hour of the infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Ethanol
Number analyzed (Participants) | 50 | 50
Participants | 22 | 24

2. Secondary Outcome: Change in Conduction Time
Description: The atrial conduction time will be measured before and after study drug infusion, and the difference between the two times will be recorded as the Change in Conduction Time
Time Frame: This will be assessed during the experimental study from the Conduction Times that are measured before and after the study drug infusion. The measurements will be performed within 1 hour of the infusion.
Measure: Median (Inter-Quartile Range); unit: ms
Arm/Group | Placebo | Ethanol
Number analyzed (Participants) | 50 | 50
ms
  Paroximal coronary sinus (CSp) to high right atrium (hRA) | 0.67 [-1.33 to 2.67] | 0.33 [-1.67 to 4.33]
  CSp to Left upper pulmonary vein (LUPV) | 3.50 [-2.00 to 12.83] | 2.88 [-3.33 to 9.17]
  Distal coronary sinus (CSd) to CSp | 0 [-1.00 to 3.00] | 0.33 [-2.00 to 2.33]
  hRA to His bundle (His) | -0.50 [-2.50 to 10.67] | -2.00 [-5.00 to 1.33]
  hRA to low right atrium (lRA) | 0.50 [-2.67 to 5.33] | 0.50 [-2.67 to 5.33]
  LUPV to right upper pulmonary vein (RUPV) | 3.67 [-9.67 to 14.83] | 3.33 [-10.00 to 11.83]
  RUPV to CSd | 1 [-6.00 to 7.67] | 2.33 [-2.33 to 10.50]
  RUPV to His | 0.33 [-6.00 to 4.67] | 4.33 [-4.00 to 11.00]

3. Secondary Outcome: Change in Atrial Effective Refractory Period (AERP)
Description: The AERP will be measured before and after study drug infusion, and the difference between the two times will be recorded as the Change in AERP
Time Frame: This will be assessed during the experimental study from the AERPs that are measured before and after the study drug infusion. The measurements will be performed within 1 hour of the infusion.
Measure: Mean (95% Confidence Interval); unit: ms
Arm/Group | Placebo | Ethanol
Number analyzed (Participants) | 50 | 50
ms | 1.59 [-4.96 to 8.14] | -3.35 [-9.89 to 3.18]

ADVERSE EVENTS:
Time Frame: 1 year post-ablation
Arm/Group | Placebo | Ethanol
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/50
Other Adverse Events (participants affected / at risk) | 1/50 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Ethanol (N=50)
Tamponade (Injury, poisoning and procedural complications) | 0 | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=50) | Ethanol (N=50)
Hypotension (General disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2017-03-30): https://cdn.clinicaltrials.gov/large-docs/43/NCT01996943/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT01996943/SAP_001.pdf